CLINICAL TRIAL: NCT00830700
Title: Telemental Health to Improve Mental Health Care and Outcomes for Children in Underserved Areas
Brief Title: Children's Attention Deficit Disorder With Hyperactivity (ADHD) Telemental Health Treatment Study
Acronym: CATTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Kathleen Myers, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12537; R01MH081997 NIMH; R01MH081997 (NIH)
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; telemental health; TMH; telepsychiatry; rural mental health services for children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CATMH intervention (Experimental): Child telemental health service delivery intervention
  Interventions: Other: CATMH intervention
- augmented TAU/PCP (No Intervention): Augmented treatment as usual with primary care physician

INTERVENTIONS:
Other: CATMH intervention — This intervention is comprised of 6-tandem-sessions of pharmacotherapy and a behavioral intervention conducted over 4-5 months. The telepsychiatrist makes prescribing decisions during the intervention following consensus guidelines for ADHD treatment. The telepsychiatrist also provides education about how neurobiological deficits of ADHD relate to observed behavioral learning and difficulties. After the 6th session, the PCP resumes care of the patient. The behavioral intervention component is delivered by therapists at each participating clinic. The therapists are trained and supervised remotely by a telepsychologist . The 6-session behavioral intervention consists of approaches to managing children's behaviors and coordination with schools and other community agencies to advocate for the child.
  Other Names: Childrens' Telemental Health Service
  Arms: CATMH intervention

SUMMARY:
While telemental health (TMH) programs are increasing nationally to address the inequity of access to psychiatric services, there are few reports of their efficacy, particularly with children. The current proposal will complete the second stage of our program development. In the first stage, we established the feasibility of a TMH service and its acceptability to families and PCPs. In the second stage of program development we will conduct a randomized clinical trial (RCT) that will determine whether it is possible to use technological advances to: 1) improve clinical outcomes for children with ADHD over outcomes achieved in usual PC; and 2) adhere to an EBT protocol implemented through TMH. Future studies will examine whether other types of complicated psychiatric disorders and EBTs are amenable to delivery via TMH.

The overall goal of this study is to determine whether an evidence-based model of care can be faithfully implemented when delivered using TMH to children with ADHD living in rural areas and can improve outcomes over treatment as usual (TAU) in PC. ADHD is an excellent focus for assessment of TMH, as PCPs encounter this disorder frequently, EBT guidelines are available, pharmacotherapy is the core treatment and is easily delivered in PC through videoconferencing, and stabilization may be readily achieved for most youth.

ELIGIBILITY:
Inclusion Criteria:

* is 5.5 - 12 years of age
* resides at home with parents/relatives
* has a dx of ADHD (CBCL DSM-oriented elevation or previous diagnosis of ADHD; C-DISC diagnosis)
* attends school 80% of time or more (including home-schooled children)
* speaks English or Spanish and parent speaks English or Spanish

Exclusion Criteria:

* child has a diagnosis of: CD, OCD, psychosis, BPD, Autism, mental retardation, major medical illness
* resident parent has a drug use problem

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 223 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Assess whether using a telemental health service delivery model effects improvement in children diagnosed with ADHD including decreased symptoms of inattention, hyperactivity, opposition and defiance and improved adaptive functioning. | baseline, 4-, 10-, 19-, and 25-weeks

SECONDARY OUTCOMES:
Assess whether using a telemental health service delivery model improves the well-being of caregivers of children diagnosed with ADHD. | baseline, 4-, 10-, 19- and 25-weeks
Assess the ability of a telemental health service delivery model to improve treatment adherence in families of children with ADHD. | baseline, 4-, 10-, 19- and 25-weeks
Assess how reliably an evidence-based treatment protocol for the treatment of children with ADHD can be implemented within a brief telemental health service. | baseline, 4-, 10-, 19-, and 25-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Myers, MD, MPH, MS, Principal Investigator — Children's Hospital and Regional Medical Center; Ann Vander Stoep, PhD, Study Director — University of Washington; Elizabeth McCauley, PhD, Study Director — University of Washington; Children's Hospital and Regional Medical Center; Wayne Katon, MD, Study Director — University of Washington; Carolyn McCarty, PhD, Study Director — University of Washington
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Derived] Rockhill CM, Carlisle LL, Qu P, Vander Stoep A, French W, Zhou C, Myers K. Primary Care Management of Children with Attention-Deficit/Hyperactivity Disorder Appears More Assertive Following Brief Psychiatric Intervention Compared with Single Session Consultation. J Child Adolesc Psychopharmacol. 2020 Jun;30(5):285-292. doi: 10.1089/cap.2020.0013. Epub 2020 Mar 11. PMID 32167784
- [Derived] Vander Stoep A, McCarty CA, Zhou C, Rockhill CM, Schoenfelder EN, Myers K. The Children's Attention-Deficit Hyperactivity Disorder Telemental Health Treatment Study: Caregiver Outcomes. J Abnorm Child Psychol. 2017 Jan;45(1):27-43. doi: 10.1007/s10802-016-0155-7. PMID 27117555
- [Derived] Rockhill CM, Tse YJ, Fesinmeyer MD, Garcia J, Myers K. Telepsychiatrists' Medication Treatment Strategies in the Children's Attention-Deficit/Hyperactivity Disorder Telemental Health Treatment Study. J Child Adolesc Psychopharmacol. 2016 Oct;26(8):662-671. doi: 10.1089/cap.2015.0017. Epub 2015 Aug 10. PMID 26258927
- [Derived] Myers K, Vander Stoep A, Zhou C, McCarty CA, Katon W. Effectiveness of a telehealth service delivery model for treating attention-deficit/hyperactivity disorder: a community-based randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2015 Apr;54(4):263-74. doi: 10.1016/j.jaac.2015.01.009. Epub 2015 Jan 29. PMID 25791143
- [Derived] Rockhill C, Violette H, Vander Stoep A, Grover S, Myers K. Caregivers' distress: youth with attention-deficit/hyperactivity disorder and comorbid disorders assessed via telemental health. J Child Adolesc Psychopharmacol. 2013 Aug;23(6):379-85. doi: 10.1089/cap.2013.0019. PMID 23952184
- [Derived] Myers K, Vander Stoep A, Lobdell C. Feasibility of conducting a randomized controlled trial of telemental health with children diagnosed with attention-deficit/hyperactivity disorder in underserved communities. J Child Adolesc Psychopharmacol. 2013 Aug;23(6):372-8. doi: 10.1089/cap.2013.0020. PMID 23952183
- [Derived] Vander Stoep A, Myers K. Methodology for conducting the children's attention-deficit hyperactivity disorder telemental health treatment study in multiple underserved communities. Clin Trials. 2013;10(6):949-58. doi: 10.1177/1740774513494880. Epub 2013 Jul 29. PMID 23897950